CLINICAL TRIAL: NCT05841186
Title: Correlation of Timing of Pegfilgrastim Administration and PIBP(Pegfilgrastim-induced Bone Pain)
Brief Title: Correlation of Timing of Pegfilgrastim Administration and PIBP.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-Q-2022-474-02
Record Dates: First submitted 2023-04-07; First posted 2023-05-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pegfilgrastim; Bone Pain; Chemotherapy; Breast Cancer; Patient-reported Outcomes; Quality of Life
Keywords: pegfilgrastim; bone pain; patient-reported outcomes; chemotherapy; Breast Cancer; health related-quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 24h group (Other): Pegfilgrastim is administrated 24 hours after completing the chemotherapy in the 24-hour group.
  Interventions: Other: Timing of pegfilgrastim administration
- 48h group (Other): Pegfilgrastim is administrated 48hours after completing the chemotherapy in the 48-hour group.
  Interventions: Other: Timing of pegfilgrastim administration
- 72h group (Other): Pegfilgrastim is administrated 72 hours after completing the chemotherapy in the 72-hour group.
  Interventions: Other: Timing of pegfilgrastim administration

INTERVENTIONS:
Other: Timing of pegfilgrastim administration — Timing of pegfilgrastim administration

SUMMARY:
According to the National Comprehensive Cancer Network (NCCN) guidelines, patients receiving high-risk or moderate-risk febrile neutropenia (FN) chemotherapy with at least one risk factor should receive prophylactic granulocyte colony-stimulating factors (G-CSFs). However, pegfilgrastim-induced bone pain (PIBP) remains a common and significant clinical issue without a satisfactory solution. Studies have reported that the incidence rate of PIBP is 71.3%, with severe bone pain occurring in 27.0% of cases. Currently, the available data on PIBP treatment are limited to case reports, reviews, and small randomized controlled trials.

The NCCN guidelines recommend preventive oral non-steroidal anti-inflammatory drugs or antihistamines as the treatment for PIBP. However, even with these preventive measures, the incidence rate of PIBP remains high at 61.1%, with severe bone pain occurring in 19.2% of cases. Severe bone pain can significantly impact the patient's health-related quality of life (HRQol), leading to potential refusal of pegfilgrastim administration and subsequent dose reduction in effective chemotherapy. Ultimately, this may have negative implications for tumor cure rates and patient survival.

Based on previous literature, it appears that delaying the administration of pegfilgrastim may be associated with a lower incidence of PIBP. Therefore, our study aims to investigate the correlation between the timing of pegfilgrastim administration and the occurrence of PIBP.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years and less than or equal to 70 years.
2. Pathologically or histologically confirmed diagnosis of primary breast cancer.
3. Able to receive the chemotherapy regimen as scheduled.
4. Able to understand Chinese and fill out the study-related questionnaires independently.
5. Given written informed consent.
6. There is no need to use prescription or over-the-counter drugs regularly because of pre-existing chronic pain.

Exclusion Criteria:

1. Suffering from bone pain due to other diseases currently.
2. Allergy or contraindication to chemotherapeutic agents or pegfilgrastim.
3. Previous use of pegfilgrastim.
4. Previous received chemotherapy.
5. Pregnancy or breastfeeding.
6. Concurrently accompanied by other primary malignant tumors.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
The area under the curve (AUC) for daily worst bone pain score for days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration) in cycle 1. | Days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration).
  Measured by Brief Pain Inventory-Short Form

SECONDARY OUTCOMES:
Incidence of bone pain | Days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration).
  Measured by Brief Pain Inventory-Short Form
Incidence of severe bone pain | Days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration).
  Measured by Brief Pain Inventory-Short Form
Duration of bone pain and severe bone pain | Days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration).
  Measured by Brief Pain Inventory-Short Form
Impact of bone pain on daily life and other aspects. | Days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration).
  Measured by Brief Pain Inventory-Short Form
Change From Baseline in European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ-C30) Score. | Before pegfilgrastim administration in the first chemotherapy cycle (baseline), day 7 after each cycle of pegfilgrastim administration.
  The EORTC QLQ-C30 is a questionnaire to assess quality of life (QoL), it is composed of 30 questions (items) resulting in 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, pain), and 6 single items (dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties). All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status indicate a better quality of life; a positive change from baseline indicates improvement. Lower scores on the symptom and single-item scales indicate a better quality of life; a negative change from baseline indicates improvement.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire Breast Cancer-23 (EORTC QLQ-BR23) Score. | Before pegfilgrastim administration in the first chemotherapy cycle (baseline), day 7 after each cycle of pegfilgrastim administration.
  The EORTC QLQ-BR23 is a questionnaire to assess quality of life (QoL), it is composed of 23 questions (items) resulting in 4 functional scales (Body Image, Future Perspective, Sexual Functioning, Sexual Enjoyment) and 4 symptom scales (Systemic Therapy Side Effects, Upset by Hair Loss, Arm Symptoms, Breast Symptoms). All of the scales measures range in score from 0 to 100. Higher score for the functioning scales indicate a better quality of life; a positive change from baseline indicates improvement. Lower scores on the symptom scales indicate a better quality of life; a negative change from baseline indicates improvement.
Change From Baseline in European Quality of Life-Five Dimension-Five Level Scale (EQ-5D-5L) Score. | Before pegfilgrastim administration in the first chemotherapy cycle (baseline), day 7 after each cycle of pegfilgrastim administration.
  The EQ-5D-5L consists of a descriptive system that defines health in terms of five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a visual analog scale (VAS) for respondents to rate their current health status from 0 (worst health) to 100 (best imaginable health). A unique EQ-5D-5L health state (or profile) for each patient was generated by combining the results for the dimensions, consisting of a five-digit code. The health states were then converted to a preference-weighted summary score (weights derived from the general population), or EQ-5D-5L health utility index, with higher scores indicating better outcomes, and a positive change from baseline indicates improvement.
Analgesic use | Days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration).
  According to the diary written by the patient about the use of the analgesic.
The area under the curve (AUC) for daily worst bone pain score for days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration) in every cycle. | Days 1 through 5 (day 1 is defined as the day of pegfilgrastim administration).
  Measured by Brief Pain Inventory-Short Form
Leukocyte count | Patients do blood routine tests on the seventh day of each chemotherapy cycle (Each cycle lasts 28 days, and day 1 denotes the day of chemotherapy completion) and when necessary.
  Measured by blood routine tests.
Incidence of febrile neutropenia | Patients monitor their oral temperature daily, and do blood routine tests on the seventh day of each chemotherapy cycle (Each cycle lasts 28 days, and day 1 denotes the day of chemotherapy completion) and when necessary.
  Measured by thermometer and blood routine tests.
Incidence of neutropenia | Patients do blood routine tests on the seventh day of each chemotherapy cycle (Each cycle lasts 28 days, and day 1 denotes the day of chemotherapy completion) and when necessary.
  Measured by blood routine tests.
Absolute neutrophil count | Patients do blood routine tests on the seventh day of each chemotherapy cycle (Each cycle lasts 28 days, and day 1 denotes the day of chemotherapy completion) and when necessary.
  Measured by blood routine tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, professor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Department of Breast Cancer, Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No